CLINICAL TRIAL: NCT00956241
Title: J-pouch Versus Side-to-end Coloanal Anastomosis After Preoperative Radiotherapy and Total Mesorectal Excision for Rectal Cancer: a Multicenter Randomized Trial
Brief Title: J-pouch Versus Side-to-end Coloanal Anastomosis After Preoperative Radiotherapy and Total Mesorectal Excision for Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Dutch Digestive Diseases Foundation (Other); Commission of Applied Clinical Research (Commissie voor Klinisch Toegepast Onderzoek: CKTO). (Unknown)
Responsible Party: A. Doeksen, MLDS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WS 01-62
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; colonic pouch; side-to-end anastomosis; preoperative radiotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- j-pouch coloanal anastomosis (Other): although a j-pouch coloanal anastomosis is a common type of anastomosis, a comparison with the side-to-end has not been made.
  Interventions: Procedure: j-pouch coloanal anastomosis
- side-to-end coloanal anastomosis (Other): in the Netherlands, the side-to-end anastomosis is the standard procedure to perform an anastomosis in case of rectal resection. therefore, the side-to-end group was our control group
  Interventions: Procedure: side-to-end coloanal anastomosis

INTERVENTIONS:
Procedure: j-pouch coloanal anastomosis
  Arms: j-pouch coloanal anastomosis
Procedure: side-to-end coloanal anastomosis
  Arms: side-to-end coloanal anastomosis

SUMMARY:
The objective of this study was to compare the functional and surgical results of the J-pouch with those of the side-to-end anastomosis and their impact on quality of life.

DETAILED DESCRIPTION:
Invalidating anorectal dysfunctions are common after restorative rectal surgery. Improvement of functional results by the technically more demanding J-pouch has been demonstrated in comparison with the straight coloanal anastomosis. In the present multicenter randomized trial we assessed whether the J-pouch is also superior to the side-to-end coloanal anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria comprised a histologically proven rectal cancer located in the middle or distal part of the rectum (≤ 10cm from the anal verge), and a WHO performance status ≤ 2.

Exclusion Criteria:

* Patients with a T1 or T4 tumor were excluded
* Patients diagnosed with distant metastases
* A medical history of colonic resection
* Anorectal surgery or chemo- radiotherapy
* Pre-existing fecal incontinence grade III or IV according to Parks10
* Life expectancy of less than one year.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2002-04; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Primary endpoint was the function of the neo-rectum as assessed by a validated functional outcome questionnaire at 4 months. | 4 months

SECONDARY OUTCOMES:
Function of the neo-rectum as assessed by the functional outcome questionnaire | 12 months
Surgical results | 4 and 12 months
Quality of life | 4 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Doeksen A, Bakx R, Vincent A, van Tets WF, Sprangers MA, Gerhards MF, Bemelman WA, van Lanschot JJ. J-pouch vs side-to-end coloanal anastomosis after preoperative radiotherapy and total mesorectal excision for rectal cancer: a multicentre randomized trial. Colorectal Dis. 2012 Jun;14(6):705-13. doi: 10.1111/j.1463-1318.2011.02725.x. PMID 21831100